CLINICAL TRIAL: NCT03064477
Title: Cost-efficacy and Acceptability of the Unified Protocol for the Treatment of Emotional Disorders in the Spanish Public Mental Health System Using a Group Format
Brief Title: The Unified Protocol for the Treatment of Emotional Disorders in Spanish Public Mental Health System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJIUP
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Emotional Disorder; Anxiety Disorders; Depressive Disorder
Keywords: Unified Protocol; Transdiagnostic approach; Public health
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All consecutive patients with emotional disorders attending any of the collaborating centers will be asked to participate in the present study. Once inclusion criteria are met, each patient will be randomly assigned to one of the two experimental groups: TAU or UP. Randomization will be performed by a researcher unrelated to the study using a computer-generated sequence (Randomizer). Randomization will be stratified according to the severity of the primary measures of depression and anxiety, using the recommended cutoff in the manuals. Stratification will be made to ensure a comparable proportion of severely depressed and anxious individuals in each group. For each subgroup (i.e., severe or less severe depression and/or anxiety), participants will be randomly assigned to the UP or to TAU.
Who Masked: Participant
Masking Description: Patients (participants) will know the treatment they have been assigned to, but they will not know whether that treatment is considered TAU or experimental (UP). Healthcare professionals and researchers will know the condition each patient has been assigned to (mandatory to provide a given type of intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (UP) (Experimental): Investigators in the present study have adapted the UP to implement it in group format in a Public Mental Health setting in Spain. This adaptation is composed of 12 treatment sessions of two hours of duration each, at a rate of one per week.
  Participants in the UP will receive UP treatment in group format instead of the usual Cognitive Behavioral Therapy in individual format. Patients in the UP condition will receive pharmacological treatment (i.e., antidepressants and / or anxiolytics) as usual.
  Interventions: Behavioral: Unified Protocol
- Treatment As Usual (TAU) (Active Comparator): Cognitive Behavioral Therapy in individual format is the treatment of choice (TAU) by psychologists and psychiatrists at the collaborating Public Mental Health Centers and Primary Care Centers, together with pharmacological treatment (i.e., antidepressants and / or anxiolytics).
  Interventions: Behavioral: Cognitive Behavioral Therapy (TAU)

INTERVENTIONS:
Behavioral: Unified Protocol — Intervention group that carries out the Unified Protocol in a group format
  Arms: Unified Protocol (UP)
Behavioral: Cognitive Behavioral Therapy (TAU) — TAU group that carries out Cognitive Behavioral Therapy in an individual format
  Arms: Treatment As Usual (TAU)

SUMMARY:
The present randomized, controlled trial will compare the cost-efficacy and acceptability of the Unified Protocol in group format against traditional individual Cognitive Behavioral Treatment in a sample of patients with emotional disorders. Ultimately, the goal of the current study is to explore whether the Unified Protocol in group format can be a cost-effective psychological intervention for emotional disorders in the Spanish National Health System, that is, one that generates long-lasting changes in symptoms, while reducing both direct and indirect economic costs associated with the treatment of emotional disorders.

DETAILED DESCRIPTION:
Emotional disorders (EDs; i.e., depressive and anxiety disorders) have become the most prevalent psychiatric disorders globally. The 12-month prevalence of anxiety and depressive disorders affect 14% and 7.8% (6.9% by major depression) of the population, respectively, and comordibity may be as high as 50%. Lifetime prevalence rates in primary care settings in Spain reveal that mood and anxiety disorders, as defined in the DSM-IV-TR, are the most prevalent psychiatric problems as well, with 35.8% and 25.6%, respectively.

As a result of their high prevalence in the population, emotional disorders have become a global health problem due to their associated costs.For instance, a study conducted in 36 countries estimated that the annual cost of treatment for depressive disorders and anxiety problems amounted to $91 billion and $56 billion, respectively. If both direct and indirect costs of these emotional disorders were accounted for, expenses increased to $925,000 million. In Spain, when both direct and indirect costs are included, mood and anxiety disorders are estimated to cost €10,763 million and €10,365 million, respectively.

Pharmacological treatment and individual cognitive behavioral therapy (CBT) are the most frequent interventions for emotional disorders in the Spanish National Health System. Therefore, increasing the efficiency of these treatments may be a way of reducing the current public health costs of emotional disorders. A recently developed form of CBT, the Unified Protocol for the Treatment of Emotional Disorders (UP), might serve the aforementioned purpose, as it can be applied to a variety of disorders simultaneously and it can be easily performed in a group format. The UP was created on the basis of the identification of common psychopathological vulnerability factors in emotional disorders, together with elements and techniques shared by disorder-specific cognitive-behavioral treatments. In the UP, traditional CBT techniques (i.e., cognitive restructuring) and contemporary practices (i.e., mindfulness) are combined to treat emotion regulation deficits, which are argued to be the underlying common factor in all emotional disorders. The UP is a structured, manual-based treatment, so it can be easily applied in a group format. This, together with the fact that the UP can be applied simultaneously to individuals with different emotional disorders, might help reduce existent waiting lists and current costs of individual treatment.

So far, studies exploring the effectiveness of the UP in a group format have led to promising findings. Overall, results suggest that the UP has between moderate and strong effect sizes on numerous outcomes, including depression, anxiety, positive and negative affect, quality of life, overall adjustment, and avoidance of negative sensations, for both anxiety and mood disorders. These studies have also revealed that between half and two thirds of patients ceased to meet diagnostic criteria after the treatment and one investigation, conducted by the investigators participating in the present study, revealed that changes remained stable 12 months after treatment completion. Despite the previous results are encouraging, conclusions should be interpreted with caution as sample sizes have been small (11 participants in two studies and 47 patients in one investigation) and cost-effectiveness of the UP in group format compared with traditional individual CBT remains unclear. Methodologically-sound, randomized, controlled trials are needed in order to replicate the aforementioned findings and to elucidate whether the UP in group format is an effective and efficient treatment option for emotional disorders in public settings.

It is expected that both interventions (CBT and UP) will be comparable in terms of effectiveness and acceptability, but treatment costs will be lower in the UP condition. To ensure the generalizability of results, the hypotheses will be tested in various public mental health centers in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety or mood disorder is the main diagnosis
* The patient is over 18 years of age
* The patient is fluent in the language in which the therapy is performed (Spanish in the present study)
* The patient is able to attend to the evaluation and treatment sessions
* The patient signs the informed consent form

Exclusion Criteria:

* The patient presents a severe mental disorder (bipolar disorder, schizophrenia, or an organic mental disorder) or there is suicide risk at the time of assessment
* The patient has used substances in the last three months (excluding cannabis, coffee, and / or nicotine)
* The patient has previously received 8 or more sessions of psychological treatment with clear and identifiable CBT principles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09-14 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the severity of depressive symptoms | Up to 12 months
  The Beck Depression Inventory-II (BDI-II) is a largely used measure that evaluates depressive symptomatology. It consists of 21 items, each including a set of four different sentences that reflect an increasing degree of depression. Responses are obtained through a 4-point Likert scale ranging from 0 (lowest degree of depressive symptomatology) to 3 (most severe symptomatology). Scores in the BDI-II range from 0 to 63. The alpha coefficient obtained in the Spanish version (.87) indicates a good internal consistency.
Change in the severity of anxiety symptoms | Up to 12 months
  The Beck Anxiety Inventory (BAI) is a frequently used measure of the severity of anxiety symptoms. The BAI includes 21 items. Each item reflects an anxiety symptom and respondents are asked to rate the extent to which the symptoms affected them during the past week. Responses are obtained through a 4-point Likert scale ranging from 0 = not at all to 3 = severely. Total score ranges from 0 to 63. The internal consistency estimate for the Spanish version of the BAI is high (.93).

SECONDARY OUTCOMES:
Change in quality of life | Up to 12 months
  The Quality of Life Index (QLI) is a self-report measure composed of 10 items, each representing a dimension of quality of life: physical disability, emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social emotional support, community and services support, personal fulfillment, spiritual fulfillment, and overall quality of life. Responses are obtained be means of a 10-point line ranging from 0 = poor to 10 = excellent. Test-retest reliability of the Spanish version of the QLI (QLI-Sp) is very good (.89).
Change in the general tendency to worry | Up to 12 months
  The Penn State Worry Questionnaire (PSWQ) was administered to patients with general anxiety disorders. It evaluates an individuals' general tendency to worry excessively. It contains 16 items that assess the intensity and frequency of preoccupation where 1 = nothing and 5 = much. The PSWQ has an excellent internal consistency (.95).
Change in obsessions and compulsions | Up to 12 months
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a semi-structured interview is used to evaluate the severity of obsessions and compulsions of patients with obsessive-compulsive disorders. It consists of 64 items, which are then grouped into 15 categories. The categories evaluate the duration, interference, discomfort, resistance, and control over obsessions and compulsions using a scale ranging from 0 = absence of symptoms to 4 = extreme severity of symptoms. The Y-BOCS has a very good internal consistency (.60-.91).
Change in the severity of panic symptoms | Up to 12 months
  The Self-reported Panic Disorder Severity Scale (PDSS-SR) evaluates the severity of symptoms in persons with panic disorders (intensity, frequency, interference, avoidance, and agoraphobic fear, among others) using a semi-structured interview. Seven Likert-type items are administered each with a 0-4 range (0 = minimum severity of symptoms and 4 = maximum severity of symptoms). The internal consistency of this instrument is good (.65).
Change in agoraphobia severity | Up to 12 months
  The Inventory for Agoraphobia (IA) examines the physiological, motor, and cognitive responses of agoraphobia patients, both when they are alone and accompanied. It consists of 69 Likert-type items. The internal consistency is high for the three subscales: physiological responses (0.94), motor responses (0.93), and cognitive responses (0.87).
Change in the severity of post-traumatic symptoms | Up to 12 months
  The Post-Traumatic Stress Disorder Symptom Severity Scale (PTSD-SSS) is used to assess the severity of symptoms in people who have experienced a traumatic life event. It contains 17 items that are classified into 3 subscales: re-experimentation, avoidance, and activation increase. The internal consistency of the scale is excellent (.92).
Change in social anxiety symptoms | Up to 12 months
  The Social interaction anxiety inventory (SIAS) is a self-reported scale assesses fear and anxiety in social interactions. It consists of 19 items that refer to the severity of symptoms, where 0 indicates nothing and 4 indicates very. The SIAS has excellent reliability estimates (.90).
Change in the severity of hypochondriacal attitudes | Up to 12 months
  The Whiteley Index of hypochondriasis (WI) consists of 14 dichotomous items, labeled yes and no, that evaluate hypochondriacal attitudes. Items are grouped into 3 subscales: bodily concern, phobia to diseases, and conviction of the presence of a disease. The internal consistency of scales in the WI is very good (.76 - .80).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Osma, Ph.D., Principal Investigator — Assistant Professor
Locations (3):
- Spain (3):
  - Hospital General Universitario de Elda, Elda
  - Clínica de Navarra, Pamplona
  - Hospital Comarcal de Vinaròs, Vinaròs

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Barlow DH, Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Allen LB, Ehrenreich-May J. Protocolo unificado para el tratamiento transdiagnóstico de los trastornos emocionales: Manual del terapeuta y manual del paciente.[The unified protocol for transdiagnostic treatment of emotional disorders: Client workbook and Therapist guide]. Madrid: Alianza Editorial; 2015.
- [Background] Beck AT, Steer R. Beck Anxiety Inventory manual. San Antonio: Psychological Corporation;1993.
- [Background] Gallagher MW, Sauer-Zavala SE, Boswell JF, Carl JR, Bullis J, Farchione TJ, Barlow DH. The Impact of the Unified Protocol for Emotional Disorders on Quality of Life. Int J Cogn Ther. 2013 Mar 1;6(1):10.1521/ijct.2013.6.1.57. doi: 10.1521/ijct.2013.6.1.57. PMID 24358405
- [Background] Osma J, Barrada JR, Garcia-Palacios A, Navarro-Haro M, Aguilar A. Internal Structure and Clinical Utility of the Anxiety Control Questionnaire-Revised (ACQ-R) Spanish Version. Span J Psychol. 2016 Oct 3;19:E63. doi: 10.1017/sjp.2016.69. PMID 27692017
- [Background] Osma J, Castellano C, Crespo E, García-PalaciosA. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in format group in a Spanish public mental health setting. PsicologíaConductual. 2015; 23 (3): 447-466.
- [Background] Carl JR, Gallagher MW, Sauer-Zavala SE, Bentley KH, Barlow DH. A preliminary investigation of the effects of the unified protocol on temperament. Compr Psychiatry. 2014 Aug;55(6):1426-34. doi: 10.1016/j.comppsych.2014.04.015. Epub 2014 Apr 27. PMID 24933653
- [Derived] Peris-Baquero O, Osma J. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Group Format in Spain: Results of a Noninferiority Randomized Controlled Trial at 15 Months after Treatment Onset. Depress Anxiety. 2023 Jun 30;2023:1981377. doi: 10.1155/2023/1981377. eCollection 2023. PMID 40224586
- [Derived] Osma J, Peris-Baquero O, Suso-Ribera C, Farchione TJ, Barlow DH. Effectiveness of the Unified Protocol for transdiagnostic treatment of emotional disorders in group format in Spain: Results from a randomized controlled trial with 6-months follow-up. Psychother Res. 2022 Mar;32(3):329-342. doi: 10.1080/10503307.2021.1939190. Epub 2021 Jun 16. PMID 34132170
- [Derived] Osma J, Suso-Ribera C, Garcia-Palacios A, Crespo-Delgado E, Robert-Flor C, Sanchez-Guerrero A, Ferreres-Galan V, Perez-Ayerra L, Malea-Fernandez A, Torres-Alfosea MA. Efficacy of the unified protocol for the treatment of emotional disorders in the Spanish public mental health system using a group format: study protocol for a multicenter, randomized, non-inferiority controlled trial. Health Qual Life Outcomes. 2018 Mar 12;16(1):46. doi: 10.1186/s12955-018-0866-2. PMID 29530035